CLINICAL TRIAL: NCT05565339
Title: PMEI Post-Market Clinical Follow-Up
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020PMEI001
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pre-existing Condition
Keywords: passive middle ear implant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Total Ossicular Replacement Prostheses:
  The primary objective for the total ossicular replacement prostheses was to achieve an ABG ≤ 20 dB by at least 25 % of the patients after the PMEI implantation
  Interventions: Device: PMEIs
- 2: Partial Ossicular Replacement Prostheses:
  The primary objective for the partial ossicular replacement prostheses was to achieve an ABG ≤ 20 dB by at least 53.8 % of the patients after the PMEI implantation.
  Interventions: Device: PMEIs
- 3: Stapesplasty Prostheses:
  The primary objective for the stapes prostheses was to achieve an ABG ≤ 20 dB by at least 86 % of the patients after the PMEI implantation.
  Interventions: Device: PMEIs

INTERVENTIONS:
Device: PMEIs — To evaluate audiological outcomes post-operatively, the air-bone gap (ABG) was assessed.
  To evaluate safety of the devices, adverse events were collected.A post-operative minimum and maximum follow-up period was not defined. The mean of the post-operative follow-up period of all patients was calculated. To assess whether implantation of PMEI affected residual hearing pre- and post-operative bone conduction thresholds were evaluated.

SUMMARY:
Confirm safety and performance of passive middle ear implants (PMEIs) in subjects with pre-existing condition which made the implantation of a MED-EL PMEI necessary

DETAILED DESCRIPTION:
Collect retrospective audiological and safety results of PMEI implanted subjects. A post-operative minimum and maximum follow-up period was not defined. The mean of the post-operative follow-up period of all patients was calculated.

ELIGIBILITY:
• Inclusion Criteria: Implanted with a MED-EL PMEI; initial implantation or revision implantation receiving a MED-EL PMEI

• Exclusion Criteria: None

Ages: 0 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population included MED-EL PMEI implanted patients with a pre-existing condition which made the implantation of a MED-EL PMEI necessary.
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
ABG | A post-operative minimum and maximum follow-up period was not defined.
  To collect post-operative PTA4 ABG results. It was expected to achieve a post-operative ABG ≤ 20 dB with a PMEI, by at least 25 % of the total ossicular replacement prostheses patients, by at least 53.8 % of the partial ossicular replacement prostheses patients, and by at least 86 % of the stapes prostheses patients.

SECONDARY OUTCOMES:
adverse events | A post-operative minimum and maximum follow-up period was not defined.
  To collect device, surgery or procedure related adverse events and bone conduction thresholds

CONTACTS AND LOCATIONS:
Locations (11):
- Austria (5):
  - Linz Kepler Universitätsklinikum GmbH, Klinik für Hals-, Nasen- und Ohrenheilkunde, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Abteilung für Hals-, Nasen- und Ohrenkrankheiten, Logopädie, Wels, Upper Austria
  - Universitätsklinikum St. Pölten, Klinische Abteilung für Hals-Nasen-Ohren, Sankt Pölten
  - Wiener Gesundheitsverbund, Klinik Landstraße, Hals-Nasen-Ohren-Allgemeine Ambulanz, Vienna
  - Universitätskliniken der MedUni Wien/AKH Wien, Universitätsklinik für Hals-, Nasen- und Ohrenkrankheiten, Vienna
- Germany (5):
  - Universitätsklinikum Erlangen, Hals-Nasen-Ohren-Klinik, Kopf- und Halschirurgie der Universität Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Freiburg, Universitätsklinik für Hals, - Nasen und Ohrenheilkunde Sektionsleitung Experimentell-klinische Otologie, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Klinik für Hals-Nasen-Ohrenheilkunde, Göttingen
  - Medizinische Hochschule Hannover, Klinik für HNO-Krankheiten, Hanover
  - Zentrum für Mittelohrchirurgie, Belegabteilung für Abteilung Hals-Nasen-Ohrenheilkunde, Lünen
- Center of Hearing and Speech Medincus, Clinical Trials Department, Nadarzyn, Kajetany, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolfram W, Zwittag PM, Niederwanger L, Rubicz N, Sprinzl G, Magele A, Beutner D, Bevis N, Schimanski E, Arndt S, Offergeld C, Arnoldner C, Riss D, Skarzynski PH, Plichta L, Hornung J, Taha L, Lenarz T, Busch S, Windisch F, Loader B. Clinical outcomes of 188 patients implanted with Med-El stapes prostheses. Eur Arch Otorhinolaryngol. 2025 Oct 15. doi: 10.1007/s00405-025-09733-x. Online ahead of print. PMID 41094222
- [Derived] Beutner D, Bevis N, Loader B, Windisch F, Arndt S, Offergeld C, Wolfram W, Niederwanger L, Zwittag PM, Rubicz N, Schimanski E, Arnoldner C, Riss D, Skarzynski PH, Plichta L, Hornung J, Taha L, Lenarz T, Busch S, Magele A, Sprinzl G. Safety and Effectiveness of the Titanium mAXIS Stapes Prosthesis: Multicentric Short-Term Outcome. Otol Neurotol. 2025 Jun 1;46(5):561-566. doi: 10.1097/MAO.0000000000004462. Epub 2025 Feb 19. PMID 40059729
- [Derived] Schimanski E, Lenarz T, Busch S, Arndt S, Offergeld C, Arnoldner C, Riss D, Hornung J, Taha L, Zwittag PM, Rubicz N, Beutner D, Bevis N, Loader B, Windisch F, Sprinzl G, Magele A, Wolfram W, Niederwanger L, Plichta L, Skarzynski PH. Safety and performance of the new med-el total ossicular replacement prostheses. Eur Arch Otorhinolaryngol. 2024 Nov;281(11):5687-5697. doi: 10.1007/s00405-024-08784-w. Epub 2024 Jul 13. PMID 39001922
- [Derived] Rasse T, Niederwanger L, Hornung J, Taha L, Arndt S, Offergeld C, Beutner D, Bevis N, Lenarz T, Teschner M, Schimanski E, Georg Sprinzl, Magele A, Skarzynski PH, Plichta L, Arnoldner C, Riss D, Loader B, Windisch F, Rubicz N, Zwittag PM. Short-term safety and effectiveness of the mCLIP partial prosthesis. Eur Arch Otorhinolaryngol. 2024 May;281(5):2353-2363. doi: 10.1007/s00405-023-08359-1. Epub 2023 Dec 22. PMID 38133806